CLINICAL TRIAL: NCT02563678
Title: Hyperbaric Oxygen, Neutrophil-oxidative Burst, and Cytokines: a Pilot Study
Brief Title: Hyperbaric Oxygen, Neutrophil-oxidative Burst, and Cytokines
Acronym: O2B
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Intermountain Health Care, Inc. (Other)
Responsible Party: Principal Investigator, Lindell Weaver, Director, Hyperbaric Medicine, Intermountain Health Care, Inc.
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 1040229
Record Dates: First submitted 2015-09-15; First posted 2015-09-30 (Estimated); Last update posted 2022-08-04 (Actual); Status verified 2022-08

CONDITIONS: Infection
MeSH Terms: conditions — Infections | interventions — Hyperbaric Oxygenation; Oxyhemoglobins

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (9):
- Diabetics with active, chronic infection (Active Comparator): Adult patients with diabetes mellitus and current antibiotic use for active infection will have blood drawn before and after their first and fourth clinical hyperbaric oxygen treatments.
  Interventions: Drug: Hyperbaric Oxygen
- No diabetes or infection (Active Comparator): Adult patients without diabetes and not using antibiotics will have blood drawn before and after their first and fourth clinical hyperbaric oxygen treatments.
  Interventions: Drug: Hyperbaric Oxygen
- Critically ill patients with infection (Active Comparator): Adult patients with acute, life-threatening infection for which hyperbaric oxygen is clinically indicated will have blood drawn before and after their first and fourth clinical hyperbaric oxygen treatments.
  Interventions: Drug: Hyperbaric Oxygen
- Carbon monoxide patients (Active Comparator): Adult patients with acute carbon monoxide poisoning will have blood drawn before and after their first clinical hyperbaric oxygen treatment.
  Interventions: Drug: Hyperbaric Oxygen
- Glucose tolerance test (Active Comparator): Diabetic patients co-enrolled in a hyperbaric oxygen and glucose control study will have blood drawn before and after their glucose tolerance test and their first clinical hyperbaric oxygen treatment.
  Interventions: Drug: Hyperbaric Oxygen
- Brain injury research subjects (Experimental): Research subjects co-enrolled in a study examining hyperbaric oxygen for post-concussive symptoms will have blood drawn before and after their first and fourth hyperbaric chamber sessions.
  Interventions: Drug: Hyperbaric Oxygen
- Hyperbaric chamber inside attendants (Experimental): Hyperbaric chamber inside attendants will have their blood drawn before, mid-session, and after their chamber exposure during their regular duty day. The hyperbaric chamber exposure will include hyperbaric air and hyperbaric oxygen components (hyperbaric air/oxygen).
  Interventions: Other: Hyperbaric Air/Oxygen
- Volunteers, hyperbaric oxygen (Active Comparator): Healthy adult volunteers will have blood drawn before and after a single hyperbaric chamber session.
  Interventions: Drug: Hyperbaric Oxygen
- Volunteers, normobaric pressure (Experimental): Healthy volunteers will have their blood drawn before and after breathing 100% oxygen at atmospheric pressure (normobaric oxygen) for 120 minutes.
  Interventions: Other: Normobaric oxygen

INTERVENTIONS:
Drug: Hyperbaric Oxygen — Hyperbaric oxygen therapy
  Other Names: HBO, HBO2
  Arms: Brain injury research subjects; Carbon monoxide patients; Critically ill patients with infection; Diabetics with active, chronic infection; Glucose tolerance test; No diabetes or infection; Volunteers, hyperbaric oxygen
Other: Hyperbaric Air/Oxygen — Breathing air inside a hyperbaric chamber, then breathing oxygen inside a hyperbaric chamber
  Arms: Hyperbaric chamber inside attendants
Other: Normobaric oxygen — Breathing 100% oxygen at normal, atmospheric pressure
  Arms: Volunteers, normobaric pressure

SUMMARY:
In this small pilot study, participants (patients and healthy volunteers) will have blood drawn before and after the study intervention (hyperbaric chamber session or normal pressure oxygen breathing. This blood will be analyzed for neutrophil oxidative burst and cytokine analysis.

DETAILED DESCRIPTION:
The investigators are interested in studying the influence of hyperbaric oxygen on neutrophils (a kind of white blood cell) and cytokines (cell proteins). Hyperbaric oxygen can enhance the way the immune system works, but the investigators don't fully know how that happens. the investigators are doing this study to learn more about this question.

ELIGIBILITY:
Cohort 1: Diabetic hyperbaric patients with active, chronic infection

Inclusion Criteria:

* Adult patients (ages 18-65) presenting for an anticipated course of at least 4 hyperbaric oxygen sessions for chronic clinical indications (possible indications include diabetic lower extremity wounds or refractory osteomyelitis)
* Diabetes mellitus
* Current antibiotic use for active infection

Exclusion Criteria:

* Prior treatment with hyperbaric oxygen within the last 30 days
* Consistent vitamin C or vitamin E supplementation in the past year
* Active tobacco use
* Pregnancy

Cohort 2: Hyperbaric patients without diabetes or active infection

Inclusion Criteria:

- Adult patients (ages 18-65) presenting for an anticipated course of at least 4 hyperbaric oxygen sessions for chronic clinical indications (possible indications include crush injury, acute peripheral arterial insufficiency, or radiation necrosis)

Exclusion Criteria:

* Prior treatment with hyperbaric oxygen within the last 30 days
* Consistent vitamin C or vitamin E supplementation in the past year
* Active tobacco use
* Pregnancy
* Diabetes mellitus
* Known or suspected viral or bacterial infection

Cohort 3: Critically ill hyperbaric patients with acute infection

Inclusion Criteria:

- Adult patients (ages 18-65) admitted to the intensive care unit for acute, life-threatening infection where hyperbaric oxygen is clinically indicated for at least 4 sessions (possible indications include gas gangrene or necrotizing fasciitis)

Exclusion Criteria:

* Prior treatment with hyperbaric oxygen within the last 30 days
* Consistent vitamin C or vitamin E supplementation in the past year
* Active tobacco use
* Pregnancy

Cohort 4:

Carbon monoxide-poisoned patients

Inclusion Criteria:

- Adult patients (ages 18-65) presenting for hyperbaric oxygen for acute carbon monoxide poisoning (up to 3 sessions)

Exclusion Criteria:

* Prior treatment with hyperbaric oxygen within the last 30 days
* Consistent vitamin C or vitamin E supplementation in the past year
* Active tobacco use
* Pregnancy
* Time interval between removal from carbon monoxide source and first hyperbaric oxygen session >12 hours

Cohort 5: Diabetic research subjects also undergoing glucose tolerance testing

Inclusion Criteria:

* Co-enrollment in glucose tolerance testing study
* Meet inclusion/exclusion profile for that study

Exclusion Criteria:

* Prior treatment with hyperbaric oxygen within the last 30 days
* Consistent vitamin C or vitamin E supplementation in the past year
* Active tobacco use

Cohort 6: Brain injury research subjects

Inclusion Criteria:

* Co-enrollment in brain injury study
* Meet inclusion/exclusion profile for that study

Exclusion Criteria:

* Known or suspected viral or bacterial infection
* Consistent vitamin C or vitamin E supplementation in the past year
* Active tobacco use

Cohort 7: Hyperbaric chamber inside attendants

Inclusion Criteria:

- Employees (ages 18-65) medically cleared to work as hyperbaric chamber inside attendants, reporting for a regular duty day

Exclusion Criteria:

* Known or suspected viral or bacterial infection
* Consistent vitamin C or vitamin E supplementation in the past year
* Active tobacco use
* Prior work in the hyperbaric chamber in the last 72 hours

Cohort 8: Healthy volunteers to receive hyperbaric oxygen

Inclusion Criteria:

* Healthy volunteers (ages 18-65)
* Medical clearance for hyperbaric oxygen exposure

Exclusion criteria:

* Hyperbaric oxygen exposure within the last 30 days
* Active chronic medical condition
* Use in the past 30 days of any over-the-counter or prescription medication or dietary supplement beyond a general multivitamin
* Active tobacco use
* History of significant health problems, including metabolic bone disease, skeletal muscle pathologies, cardiac or peripheral cardiovascular system abnormalities, clotting disorders, coronary artery disease, peripheral vascular disease, stroke, cancer, high cholesterol or triglycerides, high blood pressure, diabetes mellitus, or impaired liver/kidney function.
* Morbidly obese (body mass index > 40 kg/m2)
* Pregnancy
* Known or suspected viral or bacterial infection

Cohort 9: Healthy volunteers to breathe 100% oxygen at atmospheric pressure

Inclusion Criteria:

- Healthy volunteers (ages 18-65)

Exclusion criteria:

* Hyperbaric oxygen exposure within the last 30 days
* Active chronic medical condition
* Use in the past 30 days of any over-the-counter or prescription medication or dietary supplement beyond a general multivitamin
* Active tobacco use
* History of significant health problems, including metabolic bone disease, skeletal muscle pathologies, cardiac or peripheral cardiovascular system abnormalities, clotting disorders, coronary artery disease, peripheral vascular disease, stroke, cancer, high cholesterol or triglycerides, high blood pressure, diabetes mellitus, or impaired liver/kidney function.
* Morbidly obese (body mass index > 40 kg/m2)
* Pregnancy
* Known or suspected viral or bacterial infection

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2015-04; Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Oxidative Burst Assay | Within 30 minutes after chamber session 1

CONTACTS AND LOCATIONS:
Overall Officials: Lindell K Weaver, MD, Principal Investigator — Intermountain Health Care, Inc.
Locations (2):
- United States (2):
  - Intermountain Medical Center, Murray, Utah
  - Intermountain Healthcare, LDS Hospital, Salt Lake City, Utah